CLINICAL TRIAL: NCT06667193
Title: Cold-Water Immersion's Effects on Physical and Mental Health: a 4-Week Randomized Trial Comparing Cold Tub Versus Cold Shower
Brief Title: Cold Water Exposure's Effects on Physical and Mental Health
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Northern Colorado (Other)
Responsible Party: Principal Investigator, Laura Stewart, Professor, University of Northern Colorado
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2404058903
Record Dates: First submitted 2024-10-10; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Cold Exposure
Keywords: Cold Water Immersion; Cold Tub; Cold Shower

STUDY DESIGN:
Intervention Model Description: Parallel, randomized design, matched for biological age
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cold Tub Immersion Group (CI) (Experimental): Participants will utilize the research cold tub area (10 ºC, 4-minutes), following a standardized protocol (see intervention description).
  Interventions: Other: Cold Water Immersion (CWI) - Cold Tub Immersion (CI)
- Cold Shower Group (CS) (Experimental): Participants will utilize the research shower area (10 ºC, 4-minutes), following a standardized protocol (see intervention description).
  Interventions: Other: Cold Water Immersion (CWI) - Cold Shower (CS)
- Control Group (CO) (No Intervention): Participants will not participate in any cold water immersion.

INTERVENTIONS:
Other: Cold Water Immersion (CWI) - Cold Tub Immersion (CI) — Once thermoneutral procedures are complete, participants in the CI group will be seated in the cold tub and submerged into the water (10º C). The sternal notch of each participant will be used as the anatomical marker to mark submersion point. Participants will sit with both arms outstretched underwater with their backs not touching the sides of the tub. Participants with a shorter stature will be provided an underwater cushion to meet the submersion requirements. The 4-minute timer will begin once confirmation of the participants submersion level and posture is determined. Once completed, the participant will be instructed to slowly exit the tub and allowed to dry and change as necessary.
  Arms: Cold Tub Immersion Group (CI)
Other: Cold Water Immersion (CWI) - Cold Shower (CS) — Once thermoneutral procedures are complete, participants in the CS group will be instructed to enter the research shower area in Gunter 1610. Within the shower area, the walls of the shower will be numbered from 1 to 4, with 1 defined as facing the faucet, 2 defined as 90° to the right of side 1, 3 defined as 180° from the faucet, and 4 defined as 270° to the right or 90° C to the left from side 1. Participants will be instructed to turn 90° to the right cycling through sides 1 to 4 and then back to 1 every 15 seconds prompted by the researcher. This will allow the participant to complete three full rotations in the shower during the 4-minute intervention time. The shower faucet is modified and oriented in a way where it only produces cold water (10º C) when turned on. Once completed, the participant will be instructed to slowly exit the shower and is allowed to dry and change as necessary.
  Arms: Cold Shower Group (CS)

SUMMARY:
An interest in cold-water immersion (CWI) to elicit diverse physiological effects has been prevalent for centuries. CWI typically consists of bodily exposure to water at temperatures ranging from 5-10º C for various durations. CWI has profound cultural significance in different areas of the world, such as in Scandinavian countries, and has emerged as a popular modality for its purported health-promoting effects. Individuals on social media have repeatedly advocated for CWI as a method to improve muscular recovery, enhance sleep, and increase immune and cognitive function. Because of this, companies that specialize in cold tub production have become popularized; however, individuals who are seeking a more cost-effective option are drawn toward cold showers for their preferred method of cold exposure. Despite the scarcity of rigorous research investigating the difference in effects of cold tub versus cold shower CWI, individuals on social media promoting CWI via a shower continue to praise its comparable benefits to that of a tub. Therefore, investigations of chronic CWI (utilizing both a cold tub and a cold shower) is vital.

Thus, the purpose of the proposed study is to explore the varying effects of chronic CWI on neural and cognitive function using a cold tub and a cold shower. Further, the study aims to investigate performance measures and immune measures to create a comprehensive understanding of CWI's implications on human physiology over time. The investigators hypothesize measures relating to mental performance and health will improve after 4-weeks of CWI, and there will be no difference between tub and shower immersion groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Aged 18-45

Exclusion Criteria:

* Current holds a cold water exposure routine (≥3 sessions in the last month, consisting of ≥4 minutes per immersion)
* Currently pregnant of planning to become pregnant
* Chronic use of anti-inflammatory medication
* Prior history of chronic disease conditions: Cardiovascular Disease, Diabetes, Cancer, Raynaud's Disease, or severe/untreated anxiety or depression

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Sustained Attention to Response Task (SART) | Visit 1B (Week 1) and Visit 2B (Week 4)
  The SART is a task used to evaluate sustained attention and inhibitory control. Participants will complete the SART task on a laboratory computer. The computerized test will display 225 randomly selected numbers ranging between 1 and 9; these numbers appear in different sizes throughout the duration of the test and are displayed in white on a black screen. Participants will be instructed to respond when each number appears by pressing the space bar on the computer's keyboard while refraining from pressing the space bar when the number 3 appears. Total error score will be calculated by assessing the number of space bar presses when no key should've been pressed as well as absent presses when a key should've been pressed.
Alternate Use Task (AUT) | Visit 1B (Week 1) and Visit 2B (Week 4)
  The Alternate Use Task is used to evaluate creativity and divergent thinking. The task will be derived from the original paper version of the AUT, in which an everyday object will be randomly selected and presented to the participant, and the participant will be tasked with thinking of a possible use for the presented object. Participants will be instructed to think of novel and unique uses that would deviate from traditional uses of the presented object. Participants will be given a blank sheet of paper and be granted 2-minutes to write down as many uses as possible. In this modified version of the original test, participants will be screened for originality, fluency, and flexibility.
Piper Fatigue Scale (PFS) | Visit 1B (Week 1) and Visit 2B (Week 4)
  Participants will be asked to complete the Piper Fatigue Scale (PFS), a 27-question questionnaire that utilizes a Likert scale (1-10) to assess subdomains of behavioral, affective, sensory, and cognitive/mood attributes of fatigue. This version of the PFS is a subjective measure of fatigue using a 10-point Likert scale ranging from 0 - 10 with 0 indicating "No Distress" and 10 indicating "A Great Deal", "Mild" to "Severe", "Pleasant" to "Unpleasant", "Agreeable" to "Disagreeable", "Protective" to "Destructive", "Positive" to "Negative", "Normal" to "Abnormal", "Strong" to "Weak", "Awake" to "Sleepy", "Lively" to "Listless", "Refreshed" to "Tired", "Energetic" to "Unenergetic", "Patient" to "Impatient", "Relaxed" to "A Great Deal", "Exhilarated" to "Depressed", "Able to Concentrate" to "Unable to Concentrate", "Able to Remember" to "Unable to Remember", and "Able to Think Clearly" to "Unable to Think Clearly".
Perceived Stress Scale (PSS) | Visit 1B (Week 1) and Visit 2B (Week 4)
  Participants will be asked to complete the Perceived Stress Scale (PSS), a classic stress assessment tool used to gauge how different situations affect feelings and perceived stress. This version of the PSS is a subjective measure of stress using a 5-point Likert scale ranging from 0 - 4 with 0 indicating "Never", 1 indicating "Almost Never", 2 indicating "Sometimes", 3 indicating "Fairly Often", and 4 indicating "Very Often".
Mindful Attention Awareness Scale (MAAS) | Visit 1B (Week 1) and Visit 2B (Week 4)
  Participants will be asked to complete the Mindful Attention Awareness Scale (MAAS), a 15-item scale designed to assess the core characteristics of mindfulness. This version of the MAAS is a subjective measure of mindfulness using a 6-point Likert scale ranging from 1 - 6 with 1 indicating "Almost Always", 2 indicating "Very Frequently", 3 indicating "Somewhat Frequently", 4 indicating "Somewhat Infrequently", 5 indicating "Very Infrequently", and 6 indicating "Almost Never".
Heart Rate Variability (HRV) | Visit 1B (Week 1) and Visit 2B (Week 4)
  Heart rate variability (HRV) will be analyzed to determine the fluctuation in the time intervals between adjacent heartbeats to assess autonomic regulation of the heart. Resting HR and HRV were measured using the electrocardiograph (GE CASE Exercise Testing System Version 6.0, Chicago, Illinois). To measure HRV, the root mean square successive difference method (RMSSD) was used with the 10-second electrocardiogram reading. Based on the outcome of this assessment, participants with SDNN values below 50 ms will be classified as unhealthy, 50-100 ms will be classified as having compromised health, and above 100 ms will be classified as healthy.
Handgrip Dynamometry | Visit 1B (Week 1) and Visit 2B (Week 4)
  Isometric grip strength will be measured by a Baseline 12-0286 Electronic Smedly Hand Dynamometer (Fabrication Enterprises, White Plains, NY). To begin the test, participants will stand upright in a relaxed position; their upper extremity peak isometric grip strength will be assessed with the shoulder in 180º of flexion, elbow at full extension, and wrist and forearm in a neutral position. When prompted, participants will squeeze the device with their dominant hand, delivering a maximal effort for 3-seconds, followed by relaxation. After 30-seconds, the test is run again. Three sets will be completed for this test, and the highest value (kg) is recorded for analysis.
Pittsburgh Sleep Quality Index (PSQI) | Visit 1A (Week 1) and Visit 2A (Week 4)
  Participants will be asked to complete the Pittsburgh Sleep Quality Index (PSQI). The PSQI is a 19-question self-reported sleep quality screening tool broken up into 7 subcategories for scoring, such as subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction.
Serum Analysis - Brain-Derived Neurotrophic Factor (BDNF) | Visit 1A (Week 1) and Visit 2A (Week 4)
  Approximately 40mL of whole blood will be collected into serum separator tubes (Beckton Dickinson, East Rutherford, NJ, USA), allowed to clot for 30-minutes at room temperature, then centrifuged at 2000 RPM for 15 min. The serum will be pipetted into 1.5 mL microcentrifuge tubes (Eppendorf AG, Hamburg, Germany) and immediately stored in a -80 °C freezer. Serum concentrations of BDNF (Sigma-Aldrich, St. Louis, MO, USA) will be determined with a commercially available enzyme-linked immunosorbent assays. Microplates will be read with an ELx800 BioTek microplate reader (BioTek Instruments, Inc., Winooski, VT, USA) at the recommended wavelength of 450 nanometers.
Serum Analysis - Cortisol | Visit 1A (Week 1) and Visit 2A (Week 4)
  Approximately 40mL of whole blood will be collected into serum separator tubes (Beckton Dickinson, East Rutherford, NJ, USA), allowed to clot for 30-minutes at room temperature, then centrifuged at 2000 RPM for 15 min. The serum will be pipetted into 1.5 mL microcentrifuge tubes (Eppendorf AG, Hamburg, Germany) and immediately stored in a -80 °C freezer. Serum concentrations of cortisol (ALPCO Diagnostics, Salem, NH, USA) will be determined with a commercially available enzyme-linked immunosorbent assays. Microplates will be read with an ELx800 BioTek microplate reader (BioTek Instruments, Inc., Winooski, VT, USA) at the recommended wavelength of 450 nanometers.
Serum Analysis - Nerve Growth Factor (NGF) | Visit 1A (Week 1) and Visit 2A (Week 4)
  Approximately 40mL of whole blood will be collected into serum separator tubes (Beckton Dickinson, East Rutherford, NJ, USA), allowed to clot for 30-minutes at room temperature, then centrifuged at 2000 RPM for 15 min. The serum will be pipetted into 1.5 mL microcentrifuge tubes (Eppendorf AG, Hamburg, Germany) and immediately stored in a -80 °C freezer. Serum concentrations of NGF (RayBiotech, Norcross, GA, USA) will be determined with a commercially available enzyme-linked immunosorbent assays. Microplates will be read with an ELx800 BioTek microplate reader (BioTek Instruments, Inc., Winooski, VT, USA) at the recommended wavelength of 450 nanometers.

SECONDARY OUTCOMES:
Anthropometric Measures - Height | Visit 1A (Week 1) and Visit 2A (Week 4)
  Height will be obtained in centimeters (cm)( using a stadiometer SECA 220 (Chino, California, USA).
Anthropometric Measures - Weight | Visit 1A (Week 1) and Visit 2A (Week 4)
  Weight will be obtained in kilograms (kg) using a Detecto standing digital scale (Webb City, Missouri, USA).
Anthropometric Measures - Lean Body Mass | Visit 1A (Week 1) and Visit 2A (Week 4)
  Lean body mass (LBM) will be measured in kilograms and evaluated using air displacement plethysmography using a calibrated BOD POD (COSMED USA Inc., Concord, CA).
Anthropometric Measures - Body Fat Percentage | Visit 1A (Week 1) and Visit 2A (Week 4)
  Body fat percentage (BF%) will be measured as a percentage of estimated body fat relative to total body mass and evaluated using air displacement plethysmography using a calibrated BOD POD (COSMED USA Inc., Concord, CA).
Hydration | Visit 1A (Week 1) and Visit 2A (Week 4)
  A refractometer (Atago, Tokyo, JPN) will be used to evaluate urine specific gravity with a dehydration cutoff point set to ≥1.020 mg/dL. Dehydrated participants will be given time to hydrate. If dehydration persisted, participants will be asked to reschedule the session. After verbal compliance and hydration status are confirmed, participants will proceed with the study's procedures.
Qualitative Assessment | Visit 1A (Week 1) and Visit 2A (Week 4)
  Participants will be asked to complete a qualitative questionnaire to indicate their perceptions of cold water therapy. The purpose of this assessment is to see if participants' perceptions change throughout the study. Further, this questionnaire allows participants to provide any extra qualitative feedback to gain a comprehensive insight on their chronic CWI experience. No scale is used in this survey; however, participants are given the opportunity to report their perceptions of cold immersion using the following choices: increases energy, reduces anxiety, improves sleep, improves mental health, improves physical health, improves immune system, reduces soreness or pain, or other [text response].
Visual Analogue Scale (VAS) of Discomfort | Every water immersion visit (days 1-12; 3 days per week for 4 weeks)
  Participants will be assessed on their subjective ratings of discomfort as they acclimate to the cold exposure. During cold-water immersion visits (at the 1-minute mark of immersion, participants will be presented with the Visual Analogue Scale (VAS) of Discomfort, a modified version of a 0-10 item pain scale. This version of the VAS is a subjective measure of discomfort using a 11-point Likert scale ranging from 0 - 10 with 0 indicating "No Discomfort" and 10 indicating "Maximal Discomfort." Because there are twelve total water immersion visits (four weeks, three days per week), the VAS is used twelve times in total.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Northern Colorado, Greeley, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
We will make all study documents available by reasonable request (Laura.stewart@unco.edu) up to 3 years after data collection is complete.
Time Frame: Start: Oct 1, 2025 - Oct 1, 2028
Access Criteria: Anyone who contacts Laura.stewart@unco.edu with a reasonable request.